CLINICAL TRIAL: NCT03457909
Title: A Novel Detachable String Magnetically Controlled Capsule Endoscopy (DS-MCE) for Viewing Esophagus and Stomach
Brief Title: Detachable String Magnetically Controlled Capsule Endoscopy for Completely Viewing of Esophagus and Stomach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, associate professor, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DS-MCE-esophagus and stomach
Record Dates: First submitted 2018-02-04; First posted 2018-03-08 (Actual); Results first posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-08

CONDITIONS: Outpatients
Keywords: string; capsule endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DS-MCE (Experimental): outpatients who have esophagus symptoms will take DS-MCE and conventional endoscopy examination examination successively.
  Interventions: Device: DS-MCE

INTERVENTIONS:
Device: DS-MCE — During the DS-MCE examination,the capsule is allowed to travel down into gastric cardia,from where the string is slowly pulled to allow the capsule to view the esophagus retrogradely.

SUMMARY:
The purpose of the study is to determine the safety and feasibility of the new technique,detachable string magnetically controlled capsule endoscopy(DS-MCE)for evaluating gastric and esophagus diseases.

DETAILED DESCRIPTION:
Esophageal capsule endoscopy(ECE)provides a novel noninvasive approach to visualize the esophagus.The main drawback for the use of ECE is its unreliable transit time which often renders an inadequate visualization of the esophagus.Thus investigators have developed the detachable string magnetically controlled capsule endoscopy(DS-MCE) which can control the movement of the capsule through the string.

This study is a prospective, single-centered, self-controlled pilot study.Outpatients who have esophagus symptoms will take conventional endoscopy examination and DS-MCE successively.

ELIGIBILITY:
Inclusion Criteria:

* outpatients who have esophagus symptoms.

Exclusion Criteria:

* known or suspected complex history of gastrointestinal obstruction, stenosis or fistula.
* dysphagia or delayed gastric emptying.
* known or suspected possibility of active bleeding of digestive tract.
* a history of abdominal operation.
* pacemaker implantation and gastrointestinal pacemaker users.
* patients who are allergic to simethicone or pronase.
* pregnant women,mental patients.
* other circumstances that doctors consider inappropriate for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers or patients with suspected esophageal diseases were prospectively enrolled in Changhai Hospital from March 2018 to June 2018.
Pre-assignment Details: This study was a prospective, self-controlled, single-centered pilot study. After enrollment, each enrolled subject first underwent DS-MCE(detachable string magnetically controlled capsule endoscopy), and subsequently EGD(esophagogastroduodenoscopy) within one week.
Groups:
- DS-MCE: outpatients who have esophagus symptoms will take DS-MCE and conventional endoscopy examination examination.
  DS-MCE: During the DS-MCE examination,the capsule is allowed to travel down into gastric cardia,from where the string is slowly pulled to allow the capsule to view the esophagus retrogradely.
Period: Overall Study
Arm/Group | DS-MCE
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | DS-MCE
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 54 [28 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Separation of Capsule and String, and Complete Viewing of Esophagus and Stomach
Description: evaluate the feasibility of the novel DS-MCE examination. The successful separation of the capsule and string was evaluated by the capsule entering the stomach and and the string being pulled out.Complete viewing of esophagus and stomach was evaluated by completing the procedure from the capsule being swallowed, the esophagus observed retrograde, to the string being pulled out after separating from the capsule.This primary outcome indicated how many participatns completed the DS-MCE examination successfully.
Time Frame: up to 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | DS-MCE
Number analyzed (Participants) | 25
Participants | 25

2. Secondary Outcome: Number of DS-MCE Associated Adverse Events
Description: evaluate the safety of DS-MCE.Record any adverse event during the procedure and after the procedure.Patients will be followed up by telephone to inquire about the symptoms of abdominal distention, abdominal pain,vomiting and other discomfort. Follow up to the end of the capsule expulsion.
Time Frame: up to 2 weeks
Measure: Number; unit: adverse events
Arm/Group | DS-MCE
Number analyzed (Participants) | 25
adverse events | 0

3. Secondary Outcome: Duration of Time Capsule is Within the Esophagus
Description: time from the capsule swallowed to the capsule entering the gastric cardia to examine the stomach
Time Frame: up to 2 weeks
Measure: Median (Full Range); unit: minutes
Arm/Group | DS-MCE
Number analyzed (Participants) | 25
minutes | 6.2 [2.2 to 22.2]

4. Secondary Outcome: Z-line Visualization
Description: Z-line represents the normal esophagogastric junction where the squamous mucosa of the esophagus and columnar mucosa of the stomach meet.We can devide the Z-line into four quadrants under capsule endoscopy. Observing all the four quadrants is considered to be a complete observation of Z-line. In this study,the number of participants with at least two quadrants of Z-line visualized was used to evaluate the Z-line visulization.
Time Frame: up to 2 weeks
Measure: Number; unit: participants
Arm/Group | DS-MCE
Number analyzed (Participants) | 25
participants | 20

5. Secondary Outcome: Quality Score of Z-line Images
Description: grade (mild, moderate,and severe) of air-bubble and saliva interference on the Z-line view(0, no intraluminal gas bubble; 1, a few gas bubbles, no limitation of interpretation; 2, an increased amount of intraluminal foam/gas bubbles, moderate limitation of visibility; 3, an amount of foam/gas bubbles)
Time Frame: up to 2 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | DS-MCE
Number analyzed (Participants) | 25
score on a scale | 0.68 [0 to 1]

6. Secondary Outcome: Degree of Comfort
Description: evaluate patient's degree of comfort throughout the procedure.Patients will be asked to fill in a questionnaire to give scores about degree of comfort throughout the procedure.Overall discomfort was scored on a scale of 0 to 10 (0, no discomfort; 10, the overall discomfort of EGD).
Time Frame: up to 2 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | DS-MCE
Number analyzed (Participants) | 25
score on a scale | 0.96 [0 to 3]

ADVERSE EVENTS:
Time Frame: All patients were followed up to 2 weeks to confirm capsule excretion and any adverse events.
Description: strings and sleeves ruptured, capsule lost, asipration of the capsule，severe choking cough and death.
Arm/Group | DS-MCE
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT03457909/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT03457909/SAP_001.pdf